CLINICAL TRIAL: NCT03046550
Title: A Phase I, Double-Blind, Dose Escalation Study to Evaluate the Safety and Pharmacokinetics of NTM-1634 vs Placebo Administered Intravenously in Healthy Adults
Brief Title: Study to Evaluate Safety and PK of NTM-1634 vs Placebo Administered Intravenously in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: NTM-1634-001; 272201600009C-2-0-1 (NIH)
Record Dates: First submitted 2017-02-01; First posted 2017-02-08 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Cohort A will have 8 total subjects. 6 subjects will receive 0.33 mg/kg of NTM-1634 and 2 subjects will receive placebo.
  Interventions: Drug: NTM-1634; Drug: Placebo
- Cohort B (Experimental): Cohort B will have 8 total subjects. 6 subjects will receive 0.66 mg/kg of NTM-1634 and 2 subjects will receive placebo.
  Interventions: Drug: NTM-1634; Drug: Placebo
- Cohort C (Experimental): Cohort C will have 8 total subjects. 6 subjects will receive 1 mg/kg of NTM-1634 and 2 subjects will receive placebo.
  Interventions: Drug: NTM-1634; Drug: Placebo

INTERVENTIONS:
Drug: NTM-1634 — NTM-1634 drug product is a mixture of four human monoclonal IgG1 antibodies. Three dose cohorts (A: 0.33 mg/kg B: 0.66 mg/kg, and C: 1 mg/kg).
Drug: Placebo — placebo

SUMMARY:
This study evaluates the safety and pharmacokinetics of NTM-1634 in healthy subjects.

DETAILED DESCRIPTION:
NTM-1634 drug product is a mixture of four human monoclonal IgG1 antibodies.

This study is a randomized, double-blind, placebo controlled dose escalation study of three dose cohorts. Cohort A: 0.33mg/kg; B: 0.66mg/kg; and C: 1 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent understood and signed
2. Healthy male or healthy, non-pregnant, non-lactating female
3. Willingness to comply and be available for all protocol procedures including inpatient confinement for 36 - 48 hours
4. Age between 18 and 45 years, inclusive on the day of infusion
5. Body Mass Index (BMI) of ≥18.5 and ≤30 kg/m2
6. If the subject is female and of childbearing potential, she has a negative urine pregnancy test at screening and negative serum test within 24 hours prior to infusion

   * Note: A woman is considered of childbearing potential unless post-menopausal (≥ 1 year without menses) or surgically sterilized via bilateral oophorectomy, or hysterectomy or bilateral tubal ligation or successful Essure placement with documented confirmation test at least 3 months after the procedure.
7. If the subject is female and of childbearing potential, she agrees to practice abstinence from sexual intercourse with men or use acceptable contraception up to visit 12 of the study

   * Note: Acceptable contraception methods are restricted to effective devices (Intrauterine Contraceptive Devices , NuvaRing®)
8. The hemoglobin, platelet count, white blood cell count and absolute neutrophil count are within normal limits
9. The urine dipstick results on protein, glucose and blood are negative or trace

   * Note: Menstruating females failing inclusion criteria due to a positive blood on urine dipstick may be retested following cessation of menses.
10. Chemistry screening laboratory tests as outlined in Section 7.5.1.4 are in the normal reference range

    * Note: The following exceptions to laboratory normal reference ranges are allowed: Creatinine, Blood Urea Nitrogen (BUN), total bilirubin, AST, ALT, lipase, amylase, Prothrombin Time (PT), Partial Thromboplastin Time (PTT) below the lower limit of normal (LLN); CK less than 400mg/ml; Glucose, potassium, total protein, and alkaline phosphatase with a toxicity grade of 1 is allowable; albumin above the upper limit of normal (ULN).
    * Laboratory values that are outside the range of eligibility but are thought to be due to an acute condition or due to laboratory error may be repeated once.
    * Abnormalities in mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), mean platelet volume (MPV), and nucleated red blood cell count (NRBC CT), which are included in a complete blood count with differential, will not be exclusions.
11. Has adequate venous access for the infusion
12. The urine drug screen is negative
13. Breathalyzer test is negative
14. Available for follow-up for the duration of the study
15. Agrees not to participate in vigorous activity 72 hours prior to dosing through day 15 post dosing

Exclusion Criteria:

1. History of a chronic medical condition that would either interfere with the accurate assessment of the objectives of the study or increase the risk profile of the subject.

   * Note: Chronic medical conditions include diabetes; Asthma requiring use of medication in the year before screening; Autoimmune disorder such as lupus, Wegener's, rheumatoid arthritis, thyroid disease; Coronary artery disease; Chronic hypertension; History of malignancy except low-grade (squamous and basal cell) skin cancer thought to be cured; chronic renal, hepatic, pulmonary, or endocrine disease (except previous asthma which has required no treatment for the past year);
2. History of severe allergic reaction of any type to medications, bee stings, food, or environmental factors or hypersensitivity or reaction to immunoglobulins.

   * Note: Severe allergic reaction is defined as any of the following: anaphylaxis, urticaria, or angioedema
3. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds)
4. Clinically significant abnormal electrocardiogram at screening.

   * Note: Clinically significant abnormal ECG results include: complete left or right bundle branch block; other ventricular conduction block; 2nd degree or 3rd degree atrioventricular (AV) block; sustained ventricular arrhythmia; sustained atrial arrhythmia; two Premature Ventricular Contractions in a row; pattern of ST elevation felt consistent with cardiac ischemia; or any condition deemed clinically significant by a study investigator
5. Positive serology results for HIV, HBsAg, or HCV antibodies
6. Febrile illness with temperature ≥38°C within 7 days of dosing
7. Pregnant or breastfeeding
8. Donated blood within 56 days of enrollment
9. Known allergic reactions to any of the study product components present in the formulation or in the processing, as listed in the Investigator Brochure
10. Treatment with another investigational drug within 28 days of dosing
11. Treatment with a monoclonal antibody at any time
12. Receipt of antibody (e.g. TIG, VZIG, IVIG, IM gamma globulin) or blood transfusion within 6 months or within 5 half-lives of the specific product given
13. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
14. Use of H1 antihistamines or beta-blockers within 5 days of dosing
15. Use of any prohibited medication within 28 days prior to study entry or planned use during the study period

    * Note: Prohibited medications include immunosuppressives (except Nonsteroidal Anti-Inflammatory Drugs [NSAIDS]); immune modulators; oral corticosteroids (topical/intranasal steroids are acceptable); anti-neoplastic agents; any vaccine (licensed or investigational)
16. Previous exposure to botulinum toxin, receipt of antibodies against botulinum toxin, or previous treatment with equine antitoxin
17. Any previous injection or planned injection within 4 months after enrollment of botulinum toxin for cosmetic reasons, spastic dysphonia, torticollis, or any other reason
18. Any specific condition that in the judgment of the investigator precludes participation because it could affect subject safety
19. Plans to enroll or is already enrolled in another clinical trial* that could interfere with safety assessment of the investigational product at any time during the study period

    * Note: Includes trials that have a study intervention such as a drug, biologic, or device
20. Is a study site employee or staff

    * Note: Site employees or staff include the PIs and sub-investigators or staff who are supervised by the PI or Sub-Investigators
21. Systolic blood pressure >140mm Hg or diastolic blood pressure >90 mm Hg
22. Resting hear rate <50 or >100 beats per minute
23. Oral temperature ≥ 38°C (100.4°F)

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
The occurrence of Serious Adverse Events following administration of NTM-1634 to the final follow-up visit | 121 days
  number of SAE
The occurrence of Adverse Events from administration of NTM-1634 to Day 57 | 57 days
  number of AE
The occurrence of changes from baseline in physical examination following administration of NTM-1634 to the final follow-up visit | 121 days
  types of changes of physical exam findings
The occurrence of changes from baseline in vital signs following administration of NTM-1634 to the final follow-up visit | 121 day
  change in vital signs
The occurrence of changes from baseline in clinical safety laboratory values following administration of NTM-1634 to the final follow-up visit | 121 day
  change in lab values
The occurrence of changes from baseline in ECG parameters post administration of NTM-1634 on Day 1 (day of infusion) | 1 day
  changes in ECG parameters

SECONDARY OUTCOMES:
The assessment of Cmax for each of the four monoclonal antibodies of NTM-1634 | 121 days
  Cmax assessments
The assessment of Tmax for each of the four monoclonal antibodies of NTM-1634 | 121 days
  Tmax assessments
The assessment of AUC(0-t) for each of the four monoclonal antibodies of NTM-1634 | 121 days
  AUC(0-t) assessments
Development of human anti-human antibodies (HAHA) via blood collection at Days 1, 29, 57, 91 and 121. | Days 1, 29, 57, 91, and 121
  antibody development

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Ruff, MD, Principal Investigator — ICON Early Phase Services, LLC
Locations (1):
- ICON Early Phase Services, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No